CLINICAL TRIAL: NCT05959382
Title: Evaluation of Clinical Success of Restorations Using Different Magnification Aids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, ipek çubukçu, Ipek Cubukcu, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ipek001
Record Dates: First submitted 2023-07-16; First posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Dental Caries
Keywords: dental loupe; restoration success; FDI criteria
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: It has 4 groups in total. The treatments were carried out
  * with no magnification aid
  * with x2 loupe
  * with x5 loupe
  * with Dental operation microscope
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- with no magnification aid treatment (No Intervention): Dental caries treatment with no magnification aid
- with x2 dental loupe (Active Comparator): Dental caries treatment with x2 dental loupe
  Interventions: Device: Dental Loupe
- with x5 dental loupe (Active Comparator): Dental caries treatment with x5 dental loupe
  Interventions: Device: Dental Loupe
- with dental operation microscope (Active Comparator): Dental caries treatment with dental operation microscope
  Interventions: Device: Dental Operation Microscope

INTERVENTIONS:
Device: Dental Loupe — Magnification aid
  Arms: with x2 dental loupe; with x5 dental loupe
Device: Dental Operation Microscope — Magnification aid
  Arms: with dental operation microscope

SUMMARY:
This study aimed to investigate the effect of using a loupe and dental operating microscope with different magnifications on the success of class II direct composite restorations.

DETAILED DESCRIPTION:
A total of 130 class II, D2 deep caries teeth of 85 patients were randomly distributed to the naked eye, 3x magnification loupe, 5x magnification loupe, 8.5x magnification dental operating microscope (DOM) groups, and direct composite restorations were made with these magnification aids. carried out. Clearfil SE Bond 2 and Clearfil Majesty Posterior composite were used in all restorations. The restorations were evaluated using FDI criteria at 1,6 and 12-month periods, and restorations were scored between 1 and 5 for all criteria.

ELIGIBILITY:
Inclusion Criteria:

* Good oral and dental care of the patient,
* The need for at least 1 Class II restoration at a depth of D2 in the posterior group teeth,
* No crowding in the tooth to be restored, tooth contact and antagonist,
* The relevant tooth is vital,
* Absence of pain on percussion and palpation of the tooth.
* Absence of any pathology in the periapical tissues in radiographic evaluation,
* The patient was informed about the study and accepted the study,
* Having agreed to attend 1 month, 6 month and 12 month control sessions,
* The patient has no systemic disease,

Exclusion Criteria:

* Presence of severe periodontal disease,
* Teeth that cannot be insulated, malposed or overloaded or not loaded at all,
* Periodontal and endodontic removal of the relevant tooth is healthy,
* the patient is undergoing orthodontic treatment,
* Recording of dry mouth is set,
* Severe bruxism habit,
* Smoking

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Restoration Success using FDI Criteria | a week after dental treatment
  FDI criteria were categorized into three groups [3]: esthetic (four criteria), functional (three criteria) and biological (one criterion) parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)